CLINICAL TRIAL: NCT06279546
Title: Comparative Evaluation of Artificial Intelligence and Endoscopists´ Accuracy in Endoscopic Ultrasound for Identifying Normal Anatomical Structures: A Multi-institutional, Cross-sectional Study
Brief Title: Artificial Intelligence vs Endoscopist Identification in EUS Normal Anatomy
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Baylor Saint Luke's Medical Center (Unknown); Beth Israel Deaconess Medical Center (Other); Barra Life Medical Center, Brazil (Unknown); Hospital Clinico Universitario de Santiago (Other); Universitair Ziekenhuis Brussel (Other); Hospital Civil de Morelia, Michoacan (Unknown); ELIAS Emergency University Hospital (Other); Larkin Community Hospital (Other); Carol Davila University of Medicine and Pharmacy (Other); mdconsgroup, Guayaquil, Ecuador (Unknown)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Other Study IDs: IECED-12345
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Diseases
Keywords: EUS; AI; Gastrointestinal
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AI-based model: AIWorks-EUS Convolutional Neural Network version 2 (CNNv2) (mdconsgroup, Guayaquil, Ecuador) applied on pre-recorded videos for the detection of normal anatomical structures.
  Interventions: Diagnostic Test: Detection of structures
- Expert endoscopists: Endoscopists with >190 EUS procedures per year, including 75 pancreatobiliary and mucosal cancer staging procedures each, 40 subepithelial cases; and 50 cases of EUS-fine needle aspiration (FNA) (25 of them being pancreatic cases); following the American Society for Gastrointestinal Endoscopy (ASGE) recommendations.
  Interventions: Diagnostic Test: Detection of structures
- Non-expert endoscopists: Endoscopists with <190 EUS procedures per year, including 75 pancreatobiliary and mucosal cancer staging procedures each, 40 subepithelial cases; and 50 cases of EUS-FNA (25 of them being pancreatic cases); following the American Society for Gastrointestinal Endoscopy (ASGE) recommendations.
  Interventions: Diagnostic Test: Detection of structures

INTERVENTIONS:
Diagnostic Test: Detection of structures — Pre-recorded videos, cropped according to the different windows (mediastinal, gastric, duodenal) will be analyzed by the AIWorks-EUS model and endoscopists on different times for recognition of the different normal anatomical structures.

SUMMARY:
Endoscopic ultrasound (EUS) visual impression is operator-dependant and can hinder diagnostic accuracy, especially in less experienced endoscopists. The implementation of artificial intelligence can potentially mitigate operator dependency and interpretation variability, helping or improving the overall accuracy.

The investigators therefore aim to compare diagnostic accuracy between artificial intelligence (AI)-based model and the endoscopists when identifying normal anatomical structures in EUS-procedures.

DETAILED DESCRIPTION:
EUS is an operator dependent procedure where accuracy depends on experience and skills. Nowadays, EUS-training can be achieved by a formal fellowship training in a center for 6-24 months or an informal training through didactic sessions with a short hands-on experience. However, parameters for a correct and complete learning experience measurement are yet to be defined. The implementation of artificial intelligence on EUS can potentially mitigate the operator-dependent variable and improve diagnostic accuracy.

Therefore, detection of normal anatomical structures on a separate basis using an AI-based model, expert and non-expert endoscopists to determine where the AI would be most helpful.

The investigators aim to compare the diagnostic accuracy of the AI-based model with the endoscopists identification of normal anatomical structures in EUS procedures.

ELIGIBILITY:
Inclusion Criteria:

* Expert gastrointestinal EUS-endoscopists.
* Non-expert gastrointestinal endoscopists training for EUS.
* Patients with chronic dyspepsia without other findings.
* Patients with previous CT images or upper digestive endoscopy reporting no other findings.
* Patients requiring EUS for surveillance due to family history of pancreatic cancer without findings on MRI.

Exclusion Criteria:

* Internet connection less than 100 MBs per second.
* Patients with abnormal structures or with visible lesions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Expert and non-expert gastrointestinal EUS-endoscopists.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 5 months
  The true positive, true negative, false positive and false negative based on detection of anatomical structures according to the an external expert endoscopist as gold-standard.

SECONDARY OUTCOMES:
Interobserver agreement | 5 months
  Comparison of diagnostic accuracies between Artificial intelligence (AI)-based model and both groups (expert and non-expert endoscopists) using Fleiss Kappa.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- IECED, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han C, Nie C, Shen X, Xu T, Liu J, Ding Z, Hou X. Exploration of an effective training system for the diagnosis of pancreatobiliary diseases with EUS: A prospective study. Endosc Ultrasound. 2020 Sep-Oct;9(5):308-318. doi: 10.4103/eus.eus_47_20. PMID 32913147
- [Background] Cho CM. Training in Endoscopy: Endoscopic Ultrasound. Clin Endosc. 2017 Jul;50(4):340-344. doi: 10.5946/ce.2017.067. Epub 2017 Jul 31. PMID 28783919
- [Background] Finocchiaro M, Cortegoso Valdivia P, Hernansanz A, Marino N, Amram D, Casals A, Menciassi A, Marlicz W, Ciuti G, Koulaouzidis A. Training Simulators for Gastrointestinal Endoscopy: Current and Future Perspectives. Cancers (Basel). 2021 Mar 20;13(6):1427. doi: 10.3390/cancers13061427. PMID 33804773
- [Background] Robles-Medranda C, Baquerizo-Burgos J, Puga-Tejada M, Del Valle R, Mendez JC, Egas-Izquierdo M, Arevalo-Mora M, Cunto D, Alcivar-Vasquez J, Pitanga-Lukashok H, Tabacelia D. Development of convolutional neural network models that recognize normal anatomic structures during real-time radial-array and linear-array EUS (with videos). Gastrointest Endosc. 2024 Feb;99(2):271-279.e2. doi: 10.1016/j.gie.2023.10.028. Epub 2023 Oct 10. PMID 37827432